CLINICAL TRIAL: NCT03668106
Title: Effect of Different Sperm Processing Methods ( Swim up, Zeta, Sperm Gradient Centrifugation ) in ICSI Outcome. "A Sperm DNA Perspective"
Brief Title: Effect of Different Sperm Processing Methods in ICSI Outcome.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no fund
Sponsor: Benha University (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Saad, Ass. prof. OB & GYN, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Hawaa-4
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Sperm DNA Fragmentation

STUDY DESIGN:
Intervention Model Description: swim up technique
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: zeta technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- swim up method (Active Comparator): Measure volume using a sterile 2 mL pipet.Transfer specimen from a plastic cup to a sterile 15 mL- conical centrifuge tube. Gently mix the specimen with equal volume of Sperm Washing Media. Centrifuge the tubes at 1500 rpm for 10 minutes.Carefully aspirate the supernatant without disturbing the pellet and resuspend the pellet in 50mcm of fresh washing medium, then place layer of 0.5 ml of washing medium gently on the surface. Incubate the tubes at a 45° angle for 1 hour for swim-up in vertical rack in a 37°C incubator. After the incubation period, aspirate the entire supernatant from the round bottom tube. Aliquots of the detached sperm were analyzed by halosperm assay for DNA fragmentation another aliquots of same supernatant were used for ICSI then fertilization, division, blastulation, pregnancy and implantation rates were tabulated and statistically tested.
  Interventions: Procedure: sperm processing method
- sperm gradient centrifugation (Active Comparator): PureSperm gradients 40 % and 80 % were used for the experiment. All procedures were conducted under sterile conditions. Using a sterile pipette, 2.0 mL of the "lower layer" (80% PureSperm gradient) was transferred into a conical centrifuge tube.
  Using a new sterile pipette, 2.0 mL of the "upper layer" (40% PureSperm gradient) was gently dispensed on top of the lower layer. A liquefied semen sample was then placed on top of the upper layer and the tube was centrifuged for 20 minutes at 300g. The upper and lower layers were carefully aspirated without disturbing the pellet. Using a transfer pipette, 2-3 mL of Ham's F10 +10% HAS was added to the pellet and the resuspended pellet was centrifuged for 7 minutes at 300g. The supernatant was then removed and the pellet was suspended in a volume of 0.5 mL of Ham's F10 + FCS 10%. Aliquots of the detached sperm were dealt with like previous arm
  Interventions: Procedure: sperm processing method
- zeta method (Active Comparator): sperm samples were diluted 5 million in 1 ml. To induce a positive charge, the tube was placed inside a latex glove up to the cap and grasping the cap, the tube was rotated two or three turns and rapidly pulled out. Each tube was kept at room temperature for 1 minute to allow adherence of the charged sperm to the wall of the centrifuge tube.
  Tubes were hold by the cap to avoid grounding of the tube. After 1 minute the tubes were centrifuged at 200g for 5 minutes. Then, the medium and pellet were discarded in order to discard non adhering sperm and other cells. The surface of tube was washed by 0.2ml of Ham's F10+ FCS 10% in order to neutralize the charge on the wall of the tube and detach the adhering sperm.
  The collected medium at the bottom of each tube was repipetted and used to rinse the wall of the same tube several times to increase the number of recovered sperm . Aliquots of the detached sperm were dealt with like previous arm
  Interventions: Procedure: sperm processing method

INTERVENTIONS:
Procedure: sperm processing method — different sperm processing method for selcting most proper sperm for ICSI

SUMMARY:
A total 180 semen samples from couples diagnosed with unexplained infertility were SDF index tested , then total 120 semen samples of patients' husbands with abnormal SDF index were randomly divided and then processed by swim up, sperm gradient centrifugation and Zeta methods. SDF and ICSI outcomes are monitored after semen processing.

DETAILED DESCRIPTION:
A total 180 semen samples from couples diagnosed with unexplained infertility were SDF index tested , then total 120 semen samples of patients' husbands with abnormal SDF index were randomly divided and then processed by swim up (G1/ n=40), sperm gradient centrifugation (G2/ n=40) and Zeta (G3/ n=40) methods. SDF test was assessed by Halosperm kit, whereas sperm morphology was assessed by spermac stain according to strict criteria. Fertilization, division, blastulation, implantation and pregnancy rates will be tabulated and statistically tested.

ELIGIBILITY:
Inclusion Criteria:

* unexplained infertile couples for 2 years
* age from 20 years old to 37 years old

Exclusion Criteria:

* endometriosis cases
* uterine factors

Ages: 20 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Sperm DNA fragmentation | 30 minutes
  measure sperm integrity by halosperm assay

SECONDARY OUTCOMES:
Oocyte fertilization rate | day 1
  no. of oocytes fertilized /total no. of oocytes
Blastulation rate | day 5
  no of embryos blastulated / total no. of embryos
pregnancy rate | 15 days
  no of pregnant cases\ all no. of cases

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Saad, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided